CLINICAL TRIAL: NCT06905288
Title: Real-world Observational Study to Evaluate the Effectiveness of Secukinumab in Biologic-naive Ankylosing Spondylitis Patients in Korea
Brief Title: Real-world Study on Secukinumab Effectiveness in Biologic-naïve Ankylosing Spondylitis (AS) Patients in Korea.
Acronym: ONSET
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457HKR01
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Ankylosing Spondylitis
Keywords: Secukinumab; Ankylosing Spondylitis; Biologic Naive; Real World Study; Korea; Rheumatology; AS Research; Rheumatic Disease; Biologics; Clinical Effectiveness
MeSH Terms: conditions — Spondylitis, Ankylosing; Rheumatic Diseases | interventions — secukinumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group 1: The group will include subjects diagnosed with ankylosing spondylitis (AS) according to the modified 1984 New York criteria, who exhibit symptoms of active disease at both screening and baseline, as indicated by a BASDAI score of ≥ 4. Eligible participants must be biologic-naive, meaning they have no prior use of TNF inhibitors (TNFi), JAK inhibitors (JAKi), or IL-17 inhibitors (IL-17i). Additionally, patients must be deemed suitable for secukinumab treatment as per the labeling guidelines set by the Ministry of Food and Drug Safety. The study will focus on individuals with a time since AS diagnosis of less than 5 years, aged between 18 and 40 years.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — This is a prospective observational study. There is no treatment allocation. The decision to initiate treatment will be based solely on clinical judgement.

SUMMARY:
This is an observational study to evaluate the effectiveness and safety of secukinumab in participants with AS who have never used TNFi, JAKi, or IL-17i drugs before.

DETAILED DESCRIPTION:
This study is an observational study to evaluate the effectiveness and safety of secukinumab in patients with ankylosing spondylitis who are naive to TNFi/JAKi/IL-17i in Korea. Subjects will be recruited from 10 institutions in Korea. The enrollment period is 8 months from the initiation at the first institution and the follow-up periods are 28 weeks(±4 weeks). Data will be gathered at initial visit, 16 weeks(±4 weeks), and 28 weeks(±4 weeks).

Secukinumab is prescribed within the scope of labeling approved in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed with ankylosing spondylitis (AS), as defined by the modified 1984 New York criteria
2. Subjects who have symptoms of active disease at screening and baseline, as evidenced by BASDAI score of ≥ 4
3. Subjects who have never used TNFi, JAKi, or IL-17i drugs before
4. Patients suitable for secukinumab treatment within the scope of labeling by the Ministry of Food and Drug Safety
5. Subjects who have a time of less than 5 years since AS diagnosis
6. Subjects who are above the age of 18 years and below 40years old
7. Subjects who give informed consent form to participate in the study

Exclusion Criteria:

1. Subjects who are in a medical or psychological condition which may prevent them from participating in the study for the study period(28±4 weeks)
2. Subjects who have congenital/traumatic spinal deformities
3. Subjects currently enrolled in other clinical studies
4. Subjects who have any contraindications to secukinumab treatment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subjects are biologic-naive AS patients who are <40 years old and have a time of less than 5 years since AS diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Baseline and 28 weeks
  The BASDAI consists of 6 questions to measure the participant's symptoms and disease activity, and each question is evaluated using a numeric rating scale from 0 to 10 or a 10 cm Visual Analog Scale (VAS) with 0 being no problem and 10 being the worst problem

SECONDARY OUTCOMES:
Change from baseline in C-Reactive Protein (CRP) | Baseline, 16 and 28 weeks
  CRP is a blood test that indicates levels of inflammation
  * CRP< 5mg/L: Normal
  * CRP>=5 mg/L: High
Change from baseline in Ankylosing Spondylitis Disease Activity Score - C-Reactive Protein (ASDAS-CRP | Baseline, 16 and 28 week
  ASDAS-CRP is the score for participant's evaluation of low back pain, peripheral pain/swelling, duration of morning stiffness, disease activity, and the disease activity score of ankylosing spondylitis calculated from CRP levels. Ranges for Disease activity status are defined as follows:
  * Disease activity status <1.3: Inactive disease
  * Disease activity status 1.3-2.1: Low disease activity
  * Disease activity status 2.1-3.5: High disease activity
  * Disease activity status >3.5 (No maximum limit): Very high disease activity
Change from baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) stratified by specific variables | Baseline, 16 and 28 weeks
  The BASDAI consists of 6 questions to measure the participant's symptoms and disease activity, and each question is evaluated using a numeric rating scale from 0 to 10 or a 10 cm Visual Analog Scale (VAS) with 0 being no problem and 10 being the worst problem. Stratified by different baseline variables
Adverse events and Serious Adverse events | From baseline up to 28 weeks
  Incidence of Adverse events and Serious Adverse events

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Jinju

REFERENCES:
- [Background] Chimenti MS, Fonti GL, Conigliaro P, Sunzini F, Scrivo R, Navarini L, Triggianese P, Peluso G, Scolieri P, Caccavale R, Picchianti Diamanti A, De Martino E, Salemi S, Birra D, Altobelli A, Paroli M, Bruzzese V, Lagana B, Gremese E, Conti F, Afeltra A, Perricone R. One-year effectiveness, retention rate, and safety of secukinumab in ankylosing spondylitis and psoriatic arthritis: a real-life multicenter study. Expert Opin Biol Ther. 2020 Jul;20(7):813-821. doi: 10.1080/14712598.2020.1761957. Epub 2020 May 13. PMID 32401062
- [Background] Kiltz U, Sfikakis PP, Gaffney K, Sator PG, von Kiedrowski R, Bounas A, Gullick N, Conrad C, Rigopoulos D, Lespessailles E, Romanelli M, Ghislain PD, Brandt-Jurgens J, Rashkov R, Aassi M, Orsenigo R, Perella C, Pournara E, Gathmann S, Jagiello P, Veit J, Augustin M. Secukinumab Use in Patients with Moderate to Severe Psoriasis, Psoriatic Arthritis and Ankylosing Spondylitis in Real-World Setting in Europe: Baseline Data from SERENA Study. Adv Ther. 2020 Jun;37(6):2865-2883. doi: 10.1007/s12325-020-01352-8. Epub 2020 May 6. PMID 32378070
- [Background] Dzubur E, Khalil C, Almario CV, Noah B, Minhas D, Ishimori M, Arnold C, Park Y, Kay J, Weisman MH, Spiegel BMR. Patient Concerns and Perceptions Regarding Biologic Therapies in Ankylosing Spondylitis: Insights From a Large-Scale Survey of Social Media Platforms. Arthritis Care Res (Hoboken). 2019 Feb;71(2):323-330. doi: 10.1002/acr.23600. PMID 29781587
- [Background] Micheroli R, Tellenbach C, Scherer A, Burki K, Niederman K, Nissen MJ, Zufferey P, Exer P, Moller B, Kyburz D, Ciurea A. Effectiveness of secukinumab versus an alternative TNF inhibitor in patients with axial spondyloarthritis previously exposed to TNF inhibitors in the Swiss Clinical Quality Management cohort. Ann Rheum Dis. 2020 Sep;79(9):1203-1209. doi: 10.1136/annrheumdis-2019-215934. Epub 2020 Jun 24. PMID 32581090
- [Background] Wang R, Ward MM. Epidemiology of axial spondyloarthritis: an update. Curr Opin Rheumatol. 2018 Mar;30(2):137-143. doi: 10.1097/BOR.0000000000000475. PMID 29227352
- [Background] Mauro D, Forte G, Poddubnyy D, Ciccia F. The Role of Early Treatment in the Management of Axial Spondyloarthritis: Challenges and Opportunities. Rheumatol Ther. 2024 Feb;11(1):19-34. doi: 10.1007/s40744-023-00627-0. Epub 2023 Dec 18. PMID 38108992